CLINICAL TRIAL: NCT06697847
Title: Assessing Taste Thresholds and Scores on Standardised Mood Questionnaires in Participants Without Mood Disorders
Brief Title: Sweet Thresholds in Healthy Volunteers Study
Status: Recruiting | Type: Observational
Sponsor: Ranvier Health Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2Brsv1
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Taste Thresholds in Healthy Volunteers
Keywords: Taste thresholds; Healthy volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Adults with no mood disorder and who have not been diagnosed with or had treatment for a mood disorder in the last 6 months.

SUMMARY:
The sweet threshold (concentration of sucrose in water) at which healthy participants can detect a sweet flavour will be recorded.

DETAILED DESCRIPTION:
The sweet threshold (concentration of sucrose in water) at which healthy participants can detect a sweet flavour will be recorded by means of application on a cotton bud to the anterior third of the tongue. Solutions will be presented in a pseudo-randomised order. Mood questionnaires will be completed (to check that participants are indeed healthy). The questionnaires used will be the Patient Health Questionnaire 9 (PHQ9), Beck's Depression Inventory (BDI) and Generalised Anxiety Disorder Questionnaire 7 (GAD-7).

This data is being collected with the intention of its use for comparison with sweet thresholds established in other populations using the same method of sweet threshold estimation.

ELIGIBILITY:
Inclusion Criteria:

. Male and female adults of 18 years old and over;

* Participants without a diagnosis of major depressive disorder (MDD) / anxiety disorder;
* Participants not taking an antidepressant during the preceding 6 months
* Not suffering from significant other mental or physical illness, such as confirmed psychosis, end of life care, or any other condition assessed as significant by the Site Investigator;
* Willing and able to comply with all study-related procedures;
* Not having COVID 19 or continuing effects of COVID 19 including altered sense of taste;
* Understands the study requirements and the treatment procedures and is able to provide written informed consent.

Exclusion Criteria:

* Taking antidepressant medication currently or during the previous 6 months;
* Known or suspected hypersensitivity or intolerance to any taste testing solutions, or any of their excipients;
* A history or presence of neurological or confounding psychiatric conditions (such as stroke, traumatic brain injury, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, or schizophrenia);
* Patients with a diagnosis of chronic pain;
* Pregnancy or possibility pregnancy, or breastfeeding;
* Participants using supplements containing psychoactive herbs (for example St Johns Wort or 5-HTP (5-Hydroxytryptophan, also known as oxitriptan);
* Participants regularly using psychoactive stimulants (for example MDMA);
* Participants unable or unwilling to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults without mood questionnaires recruited by word of mouth and posters in retail establishments in England and Wales
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-27 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-14 (Estimated)

PRIMARY OUTCOMES:
Sweet taste threshold | From enrolment to a final taste test 6 weeks later
  Sweet taste threshold established by applying varying concentrations of sucrose solution to the tongue and assessing whether a sweet taste can be detected by the participant. The sweet threshold is the minimum concentration at which a participant can reliably detect the sweet flavour.

SECONDARY OUTCOMES:
Score on Becks Depression Inventory | From enrolment to a final questionnaire 6 weeks later
  Becks depression inventory will be completed by the participant at the first and last visit. The score will be calculated to check that the participant is free of mood disorder. The scale ranges from 1-40 and a score of less than 10 is normal. Higher scores suggest increasing degrees of depression.
Score on Patient Health Questionnaire 9 | From enrolment to a final questionnaire 6 weeks later
  Patient Health Questionnaire 9 will be completed by the participant at the first and last visit. The score will be calculated to check that the participant is free of mood disorder. The scale ranges from 0-27 and a score less than 5 suggests the subject is not depressed.
Score on Generalised Anxiety Disorder scale 7 | From enrolment to a final questionnaire 6 weeks later
  Generalised Anxiety Disorder scale 7 will be completed by the participant at the first and last visit. The score will be calculated to check that the participant is free of mood disorder. The scale ranges from 0-21. A score of less than 4 suggests minimal anxiety and increasing scores suggest greater anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Westbury Lodge, Westbury Park, Bristol, City Of Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data collected contains sensitive information and even when anonymised contains commercially sensitive information